CLINICAL TRIAL: NCT01215929
Title: Amphetamine Withdrawal Paradigm in Humans
Brief Title: Studying Amphetamine Withdrawal in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110743
Record Dates: First submitted 2010-10-01; First posted 2010-10-07 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine withdrawal; mood; retention; sleep
MeSH Terms: interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextroamphetamine (Active Comparator)
  Interventions: Drug: Dextroamphetamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextroamphetamine — Thirty treatment-seeking methamphetamine dependent volunteers will be admitted to a residential facility and be inducted onto d-amphetamine during week 1 of the study. 15 Participants then will be randomized by severity of methamphetamine dependence, sex, amphetamine withdrawal questionnaire score and history of Attention Deficit Hyperactivity Disorder to receive oral d-amphetamine at a dose of 30 mg twice daily for 2 weeks.
  Arms: Dextroamphetamine
Drug: Placebo — Thirty treatment-seeking methamphetamine dependent volunteers will be admitted to a residential facility in this 4-week, double-blind, placebo-controlled, clinical trial and be inducted onto d-amphetamine during week 1 of the study. 15 Participants then will be randomized by severity of methamphetamine dependence, sex, amphetamine withdrawal questionnaire score and history of Attention Deficit Hyperactivity Disorder to receive oral placebo tablets twice daily for 2 week.
  Arms: Placebo

SUMMARY:
Methamphetamine use is very common in the US and is associated with serious medical and psychiatric problems. There has also been a significant increase in the number of patients entering treatment for methamphetamine dependence, however, no pharmacologic treatment has been identified as effective in treating methamphetamine addiction. Given that withdrawal from methamphetamine is thought to contribute to relapse to methamphetamine use during early treatment, it is important to examine potential pharmacologic agents for alleviating withdrawal. Thus, this study is designed to study methamphetamine withdrawal in humans. To this end, 30 methamphetamine dependent participants (ages 18-65 years) will be entered into a 4-week residential study. Urine samples will be obtained at baseline to ensure recent methamphetamine use. Intake assessments will include cognitive testing, standardized assessment of depression and anxiety, profile of mood states, methamphetamine selective severity assessment, methamphetamine withdrawal assessment, sleep quality and quantity, a pre-attentional measure and attentional measure. Upon admission to the residential facility, all study participants will be started on (20-30mg) long acting amphetamine/d-amphetamine and stabilized over the first 5 days. After stabilization participants will be randomized based on sex, amphetamine withdrawal questionnaire score, and methamphetamine selective severity assessment score to either continued treatment with amphetamine/d-amphetamine or placebo for 2 weeks. All subjects will then be placed on placebo for the last 7 days. The investigators hypothesis is that stopping amphetamine administration in methamphetamine dependent individuals will negatively impact mood, sleep and cognitive function in a time-limited fashion that may differ depending upon the measure and that attentional, but not pre-attentional, measures will be adversely affected in those receiving placebo compared to those maintained on amphetamine.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old
* not currently enrolled in a treatment program
* history of methamphetamine use with recent use confirmed by a positive urine toxicology screen for amphetamines during the month prior to study entry
* self-reported Methamphetamine use on at least 15 of the past 30 days
* use of at least one half gram of methamphetamine per week during the month prior to study entry
* women of childbearing age must have a negative pregnancy test to enroll in this study

Exclusion Criteria:

* current diagnosis of alcohol, opiate, or sedative physical dependence
* ill health (e.g., major cardiovascular, renal, endocrine, hepatic disorder)
* history of schizophrenia, or bipolar type I disorder
* present or recent use of over-the-counter or prescription psychoactive drug or drug(s) that would be expected to have major interaction with d-amphetamine
* medical contraindication to receiving study medications (e.g., previous adverse reaction to d-amphetamine)
* chronic pain condition (due to impact on neurophysiological responses
* current suicidality or psychosis
* liver function tests (i.e., liver enzymes) greater than three times normal levels
* pregnancy or breastfeeding
* children 18-20 will be excluded because the P50 potential is not fully developed in children and adolescents

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical SCiences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dextroamphetamine: Dextroamphetamine: Thirty-five treatment-seeking methamphetamine dependent volunteers were admitted to a residential facility and inducted onto d-amphetamine during week 1 of the study. 18 Participants were be randomized by severity of methamphetamine dependence, sex, amphetamine withdrawal questionnaire score and history of Attention Deficit Hyperactivity Disorder to receive oral d-amphetamine at a dose of 30 mg twice daily for 2 weeks.
- Placebo: Placebo: Thirty-four treatment-seeking methamphetamine dependent volunteers will be admitted to a residential facility in this 4-week, double-blind, placebo-controlled, clinical trial and be inducted onto d-amphetamine during week 1 of the study. 17 Participants were randomized by severity of methamphetamine dependence, sex, amphetamine withdrawal questionnaire score and history of Attention Deficit Hyperactivity Disorder to receive oral placebo tablets twice daily for 2 weeks.
Period: Overall Study
Arm/Group | Dextroamphetamine | Placebo
Started | 18 | 17
Completed | 12 | 12
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dextroamphetamine | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.00 (9.76) | 33.67 (6.34) | 35.36 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Measure of Methamphetamine Withdrawal
Description: Total score on the Methamphetamine Withdrawal Assessment scale (MAWA) based on DSMIV criteria for amphetamine withdrawal. This questionnaire is comprised of 13 items which describe symptoms associated with the cessation of chronic amphetamine use for which participants indicate severity on a 4-point scale. The minimum score indicating no methamphetamine withdrawal symptoms is 0 and the maximum score is 4 indicating that a patient has the most severe withdrawal symptom related to that question. The subscales are the 13 questions and the total score is the sum of all the scores for the 13 items on the scale. The range minium and better outcome is a lower score. The range is from 0-52. The worse outcome is reflected in a higher score.
Time Frame: at the end of week 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo: Thirty-five treatment-seeking methamphetamine dependent volunteers will be admitted to a residential facility in this 4-week, double-blind, placebo-controlled, clinical trial and be inducted onto d-amphetamine during week 1 of the study. 17 Participants were randomized by severity of methamphetamine dependence, sex, amphetamine withdrawal questionnaire score and history of Attention Deficit Hyperactivity Disorder to receive oral placebo tablets twice daily for 2 weeks.
Arm/Group | Dextroamphetamine | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 3.7283 (3.37) | 10.056 (3.45)

ADVERSE EVENTS:
Arm/Group | Dextroamphetamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 8/18 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dextroamphetamine (N=18) | Placebo (N=17)
Insomnia (Psychiatric disorders) | 3 | 2
Headache (Nervous system disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes